CLINICAL TRIAL: NCT05821322
Title: Evaluating the Appropriate Blood Glucose Target Before and During Moderate Intensity Aerobic Exercise in Adults With Type 1 Diabetes Using Do-it-yourself Automated Insulin Delivery (AID) Systems (the GUARDIA [GlUcose tARget DIY-AID] Trial)"
Brief Title: Blood Glucose Target Before and During Exercise in Adults With Type 1 Diabetes Using an Artificial Pancreas
Acronym: GUARDIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: University of Alberta (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Professor of Medicine, Director, Research Platform on Obesity, Metabolism and Diabetes, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2023-1223
Record Dates: First submitted 2023-03-20; First posted 2023-04-20 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes
Keywords: Artificial pancreas; Exercice; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Temporary target of 8.3 mmol/L (Active Comparator): Current commercial artificial pancreas thresholds. Temporary target set 60 minutes before the intervention.
  Interventions: Other: Physical activity trial intervention
- Temporary target of 8.8 mmol/L (Experimental): Temporary target set 60 minutes before the intervention
  Interventions: Other: Physical activity trial intervention
- Temporary target of 9.3 mmol/L (Experimental): Temporary target set 60 minutes before the intervention
  Interventions: Other: Physical activity trial intervention

INTERVENTIONS:
Other: Physical activity trial intervention — 60 minutes aerobic ergocyle exercice at 60% VO2 Peak

SUMMARY:
Despite major technological advances in type 1 diabetes (artificial pancreas), the management of hypoglycemia remains a major challenge, especially during and after physical activity. The primary outcome is to determine the temporary blood glucose (BG) target to be set 60 minutes before aerobic exercise in people with type 1 diabetes (PWT1D) using do-it-yourself automated insulin delivery (DIY-AID) systems. Three glycemic thresholds to be applied 60 minutes before physical activity will be tested in 32 people on AID-DIY: 8.3 (current target for commercial AID systems), 8.8, and 9.3 mmol/L. Each participant will perform 3 sessions of moderate aerobic physical activity (ergocycle) at 60% of vo2peak with a different glycemic target each time (random order). Plasma glucose will be measured every 20 minutes before and during physical activity, and blood glucose measured by continuous glucose reading (DEXCOM) for 24 hours post-intervention. Once the best glycemic target is selected, participants could come to the research center for 1 or 2 more voluntary interventions to test the threshold during 1) fasting exercise and 2) late luteal phase of the menstrual cycle.

DETAILED DESCRIPTION:
This study follows a randomized, cross-over design and aims to test tree temporary BG targets (8.3, 8.8 and 9.3 mmol/L), resulting in 3 intervention visits per participants. A total of 32 participants will be recruited and randomized for this study.

Intervention visit:

* Participants will be admitted at the research center (IRCM; Montréal or Alberta) at 15:30.
* A venous catheter will be installed for plasma glucose and insulin measurements.
* At 16:00, the temporary BG target will be set in the DIY-AID system and blood sampling will begin.
* At 16:40, if glucose is < 5.5 mmol/L, 16g carbohydrate (CHO; 4 Dex4®) will be provided.
* At 16:55, a smaller sample will be taken only to verify glucose level. If glucose is < 5.5 mmol/L, 16g CHO (4 Dex4®) will be provided and exercise start will be postponed by at least 15 minutes or until glucose level is > 5.5 mmol/L. If more than three CHO intake are needed, the test will be canceled and rescheduled.
* At 17:00, exercise will be started if glucose is > 5.5 mmol/L. The exercise will consist of 60 minutes on the ergocycle at 60% of pre-determined VO2peak (moderate intensity).
* At 18:00, exercise and temporary BG target will be stopped. Blood sampling will continue for 1-hr during recovery.
* At 19:00, participant will be discharged. If glucose level is below 5.0 mmol/L, a snack of 16g CHO (4 Dex4®) will be offered. Participants will have the option to bring their dinner and eat it at the research facility before leaving if they prefer.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18 and 65 years old.
* Clinical diagnosis of type 1 diabetes for 1 year. (Note: The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not needed.)
* Treatment using DIY-AID system for 3 months.
* Own a smartphone or tablet to use the mobile application: Keenoa, Fitbit App
* Using Dexcom G6 and willing to share CGM data with the research team.
* Using rapid- (e.g., Aspart, Lispro or Glulisine) or ultra-rapid (e.g., FiAsp) acting insulin analogs.
* HbA1c < 8.5%.

Exclusion Criteria:

* Major complication within the previous 3 months (e.g., severe hypoglycemia requiring assistance, diabetic ketoacidosis, or cardiovascular event).
* Restriction in PA due to significant diabetes complications (e.g., severe peripheral neuropathy, active proliferative retinopathy, etc.) or other type of limitations (e.g., orthopedic, severe arthritis, etc.). Uncontrolled hypertension (e.g., blood pressure > 150 mmHg systolic or > 95 mmHg diastolic).
* Ongoing pregnancy or breastfeeding.
* Inability to give consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma glucose during exercise | 60 minutes (during exercice)
  To determine the temporary blood glucose (BG) target to be set 60 minutes before aerobic exercise in PWT1D using DIY-AID systems which will be associated with the smallest change in glucose during exercise by testing the targets of 8.3 (current target for commercial AID systems), 8.8, and 9.3 mmol/L.

SECONDARY OUTCOMES:
Time in range during exercice: menstrual cycle phases | 60 minutes (during exercice)
  Volunteer participants will return in the luteal phase of the menstrual cycle to repeat the intervention at the glycemic threshold targeted during the primary outcome.
Time in range (during fasting exercice) | 60 minutes (during exercice)
  The intervention will be repeated at the glycemic threshold targeted during the primary outcome
Number of hypoglycemic episodes | 60 minutes (during exercice)
  number of hypoglycemic episodes (plasma glucose < 4.0 mmol/L) during exercise.
Number of participants who required oral treatment during exercise | 60 minutes (during exercice)
  Number of participants who required oral treatment during exercise for: a) plasma glucose value < 4.5 mmol/L and b) plasma glucose value < 4.0 mmol/L.
Lowest plasma glucose | 60 minutes (during exercice)
  Lowest plasma glucose level during exercise
Plasma glucose at 60 minutes | 60 minutes
  plasma glucose level at the end of exercise
Carbohydrate consumption (g) | 60 minutes (during exercice)
  amount of carbohydrate (CHO) needed to increase glucose value
Insulin on board (units) | 60 minutes (during exercice)
  Insulin on board or active insulin at exercise onset (Units will be collected on insulin pump) from start to finish
Plasma insulin | 60 minutes (during exercice)
  plasma insulin changes from exercise start to finish (uU/mL)
Percent time in range, in hypoglycemia and in hyperglycemia | 6 hours post-exercice
  Percentage of time < 3.0 mmol/L, between 3.0-3.9 mmol/L, between 3.9-10.0 mmol/L, between 10.1-13.9 mmol/L, and > 13.9 mmol/L post-exercice until 6 am
Percent time in range, in hypoglycemia and in hyperglycemia | midnight to 6 am
  Percentage of time < 3.0 mmol/L, between 3.0-3.9 mmol/L, between 3.9-10.0 mmol/L, between 10.1-13.9 mmol/L, and > 13.9 mmol/L post-exercice until 6 am
Mean CGM glucose | 24 hours post-exercice
  post-exercice until 6 am
Glucose variability | midnight to 6 am
  post-exercice until 6 am; assessed by the CGM standard deviation
Coefficient of variation | midnight to 6 am
  post-exercice until 6 am; assessed by the coefficient of variation
Coefficient of variation | 24 hours post-exercice
  post-exercice until 6 am; assessed by the coefficient of variation
Glucose variability | 24 hours post-exercice
  post-exercice until 6 am; assessed by the CGM standard deviation
Number of participants requiring an oral treatment for hypoglycemia | midnight to 6 am
  Number of participants requiring an oral treatment for hypoglycemia (< 3.9 mmol/L) until 6 am.
Number of participants requiring an oral treatment for hypoglycemia | 24 hours post-exercice
  Number of participants requiring an oral treatment for hypoglycemia (< 3.9 mmol/L) until 6 am.
Hypoglycemia with treatment | 24 hours post-exercice
  Total number of hypoglycemia episodes requiring treatment
Hypoglycemia with treatment | midnight to 6 am
  Total number of hypoglycemia episodes requiring treatment
Carbohydrate needed (g) | midnight to 6 am
  total amount of carbohydrate (CHO) needed to treat hypoglycemic events.
Carbohydrate needed (g) | 24 hours post-exercice
  total amount of carbohydrate (CHO) needed to treat hypoglycemic events.

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, MD, PhD, Principal Investigator — IRCM
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No